CLINICAL TRIAL: NCT02725372
Title: A Phase 3, Placebo Controlled, Double-Blind, Randomized, Clinical Study to Determine Efficacy, Safety, and Tolerability of Pulsed, Inhaled Nitric Oxide (iNO) Versus Placebo in Symptomatic Subjects With PAH (Part 1 and Part 2)
Brief Title: Clinical Study of Pulsed, Inhaled Nitric Oxide Versus Placebo in Symptomatic Subjects With PAH
Acronym: INOvation-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial stopped for futility
Sponsor: Bellerophon Pulse Technologies (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULSE-PAH-004
Record Dates: First submitted 2016-01-19; First posted 2016-04-01 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; Inhaled Nitric Oxide; iNO; long term oxygen therapy; oxygen therapy
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide 75mcg/KgIBW/Hr (Experimental): Part 1:
  15Mcg/kg IBW/hr during Run-in Period dose titrated to Inhaled Nitric Oxide / 75mcg/KgIBW/Hr upon randomization to treatment arm.
  Part 2: iNO 75 mcg/kg IBW/hr Open Label Treatment (Open Label Treatment - All Subjects)
  Interventions: Drug: Inhaled Nitric Oxide 75 mcg/kg IBW/hr
- Placebo (Placebo Comparator): Part 1:
  Placebo dose setting 15mcg/kg IBW/hr Run In Period / Placebo dose setting 75 mcg/kg IBW/hr treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide 75 mcg/kg IBW/hr — Inhaled Nitric Oxide 15mcg/Kg IBW/hr for two week run in period dose titrated to Inhaled Nitric Oxide 75 mcg/kg IBW/hr at randomizationTreatment Period (Week 3 to Week 18)
  Other Names: Inhaled Nitric Oxide; iNO
  Arms: Inhaled Nitric Oxide 75mcg/KgIBW/Hr
Drug: Placebo — Part 1 Placebo arm: Inhaled Nitric Oxide 15mcg/Kg IBW/hrfor two week run in period dose titrated to Inhaled Nitric Oxide 75 mcg/kg IBW/hr at randomizationTreatment Period
  Other Names: Inhaled Nitric Oxide; iNO
  Arms: Placebo

SUMMARY:
Phase 3, placebo controlled, double-blind, randomized clinical study to determine safety, tolerability, and efficacy of pulsed, inhaled nitric oxide (iNO) versus placebo in symptomatic subjects with pulmonary arterial hypertension (PAH). Part 1 and Part 2

DETAILED DESCRIPTION:
Phase 3, placebo controlled, double-blind, randomized, clinical study to determine safety, tolerability and efficacy of pulsed inhaled nitric oxide (iNO) versus placebo as add-on therapy in subjects with pulmonary arterial hypertension (PAH) who remain symptomatic on approved PAH monotherapy or combination approved PAH therapy and long term oxygen therapy (LTOT). (Part 1 and Part 2)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (and assent as appropriate) prior to the initiation of any study mandated procedures or assessments
2. A confirmed diagnosis of PAH Group 1 who have either idiopathic PAH (IPAH), heritable PAH, drug and toxin-induced PAH, associated PAH (APAH) with connective tissue disease (CTD), APAH with repaired simple congenital systemic to pulmonary shunt (i.e., atrial septal defect, ventricular septal defect and/or patent ductus arteriosus; complete repair at least 1 year prior to Screening), APAH with human immunodeficiency virus (HIV), or APAH with portal hypertension
3. Subjects receiving at least one PAH specific therapy (ERA or PDE-5 inhibitor, or inhaled, subcutaneous, or intravenous prostacyclin or a prostacyclin analog) with the same type of therapy for at least 3 months with stable dosing 4 weeks prior to Screening. (Subjects should be receiving optimal therapy according to the disease severity)
4. Subjects using oxygen therapy by nasal cannula for at least 4 weeks prior to Screening
5. PAH diagnosis confirmed by RHC within the previous 5 years, according to the following definitions:

   * PVR ≥ 400 dynes.sec.cm-5 (5 Wood units)
   * mPAP ≥ 25 mmHg
   * PCWP or LVEDP ≤ 15 mmHg
   * Subjects who otherwise meet all the inclusion criteria and none of the exclusion criteria but have not undergone a RHC within the previous 5 years may be considered eligible for the study if they undergo a RHC and then meet the pulmonary hemodynamics criterion
6. 6MWD ≥ 100 meters and ≤ 450 meters prior to randomization
7. WHO Functional Class II-IV. Subjects with WHO Functional Class IV should be treated with prostacyclin or a prostacyclin analog (subcutaneous or intravenous), plus at least one additional PAH specific therapy (ERA or PDE-5), if available to the subject and reimbursed by health insurance
8. Age between 18 and 85 years (inclusive)
9. Willingness to use INOpulse delivery device for at least 12 hours per day
10. Willingness to continue on study drug until the subject has completed Week 18 assessments
11. Female subjects of childbearing potential must have a negative pre-treatment pregnancy test (serum or urine). All female subjects should take adequate precaution to avoid pregnancy.

Exclusion Criteria:

1. Subjects with known HIV infection who have a history within the past 3 months of any opportunistic pulmonary disease (e.g., tuberculosis, Pneumocystis carinii pneumonia, or other pneumonias) at the time of Screening 2. PAH associated with untreated thyroid disorders, glycogen storage disease, Gaucher's disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders or splenectomy 3. Subjects with pulmonary conditions that may contribute to PAH including, but not limited to, chronic bronchiectasis, cystic fibrosis, or other pulmonary condition that the Investigator may deem to contribute to the severity of the disease or impair the delivery of iNO due to airway disease 4. Subjects receiving riociguat 5. Subjects receiving oral prostanoids as monotherapy 7. PAH associated with significant venous or capillary involvement, known or suspected pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis 8. Any subject with WHO PH Groups 2, 3, 4 or 5 9. Subjects with any of the following cardiac abnormalities:

a. Underlying cardiomyopathy or clinically significant aortic or mitral valve disease in the opinion of the investigator b. Left ventricular systolic dysfunction (LVSD), i.e., left ventricular ejection fraction (LVEF) < 40% or left ventricular shortening fraction (LVSF) < 22%, as determined by local reading c. Current symptomatic coronary artery disease, myocardial infarction within 1 year, or any coronary artery interventions within 6 months 10. Systemic hypertension defined as systolic blood pressure (SBP) > 160 mmHg and/or diastolic blood pressure (DBP) > 100 mmHg persistent at Screening after a period of rest (treated or untreated) 11. Subjects with a history of deep vein thrombosis, pulmonary embolism/infarction or prothrombotic disorder must have had chronic thromboembolic pulmonary hypertension (CTEPH) excluded by ventilation/perfusion lung (V/Q) scan 12. Severe obstructive lung disease defined as both a forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 55% of predicted value 13. Moderate to severe restrictive lung disease: total lung capacity (TLC) < 60% of predicted; if TLC 60% to 70% predicted, a high resolution CT scan showing diffuse disease or more than mild patchy disease 14. Any subject who develops or has developed a PCWP > 20 mmHg during acute vasodilator testing (AVT) 15. Systemic hypotension defined as SBP < 90 mmHg persistent at Screening after a period of rest 16. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C 17. On dialysis 18. Acute or chronic physical impairment (other than dyspnea due to PAH) that would limit the ability to comply with study procedures or adherence to therapy (i.e., 6MWT), including carrying and wearing the pulsed delivery device per study protocol, or medical problem(s) likely to preclude completion of the study 19. Pregnant or breastfeeding females at Screening 20. Administered L-arginine within 1 month prior to Screening 21. Known concomitant life-threatening disease with a life expectancy less than 1 year 22. Atrial septostomy within 3 months preceding randomization 23. The concurrent use of the INOpulse device with a continuous positive airway pressure (CPAP), Bilevel positive airway presure BiPAP, or any other positive pressure device.

24. Use of investigational drugs or devices within 1 month prior to Screening (other than acute vasodilator testing with iNO) 25. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study 26. Any subject who has been enrolled in any previous clinical study with inhaled NO administered through pulse delivery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (109):
- United States (37):
  - Arizona Pulmonary Specialists, Ltd, Phoenix, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - UC San Diego / Pulmonary, Critical Care and Sleep Medicine Division, La Jolla, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - Pulmonary Disease Specialists, PA, Kissimmee, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Pulmonary and Critical Care of Atlanta, Atlanta, Georgia
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - Wellstar Medical Group - Pulmonary Medicine, Marietta, Georgia
  - Bluhm Cardiovascular Institute, Clinical Trials Unit, Chicago, Illinois
  - HeartCare Midwest, Peoria, Illinois
  - Kentuckiana Pulmonary Associates (KPA), Inc. - Louisville, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - New York Presbyterian Brooklyn Methodist Hospital - Division of Pulmonary/Critical Care/Sleep, Brooklyn, New York
  - Winthrop University Hospital, Clinical Trials Center, Mineola, New York
  - NYU Medical Center, Division Pulmonary, Critical Care and Sleep Medicine, New York, New York
  - Montefiore Medical Center - Weiler Division, The Bronx, New York
  - University of Cincinnati Medical Ctr, Dept of Internal Medicine / Pulmonary, Critical Care & Sleep Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Legacy Medical Group - Pulmonary Clinic, Portland, Oregon
  - The Oregon Clinic, PC, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - MedTrial, LLC, Columbia, South Carolina
  - Sioux Falls Cardiovascular, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center of Dallas, Dallas, Texas
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - St Vincent's Public Hospital, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
- Austria (2):
  - Innsbruck Medical University, University Hospital for Internal Medicine VI, Pneumology, Innsbruck, Tyrol
  - AKH-Vienna, Medical University of Vienna, Vienna
- Belgium (2):
  - Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg -, Leuven, Brabant
  - Hopital Erasme - Service de Cardiologie, Brussels
- Canada (3):
  - Faculty of Medicine / Peter Lougheed Center / Respiratory Research, Calgary, Alberta
  - Lawson Clinical Research Services / London Health Sciences Centre - VH, London, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
- Fundación Abood Shaio, Bogotá, Bogota D.C., Colombia
- University Hospital centre Zagreb, Zagreb, Croatia
- Vseobecna Fakultni Nemocnice v Praze (VFN), Prague, Bohemia, Czechia
- France (5):
  - Centre Hospitalier Universitaire (CHU) Hopitaux de Rouen - Hopital Charles Nicolle, Rouen, Normandy
  - Centre Hospitalier Universitaire de Grenoble (CHU Grenoble) - Clinique de Pneumologie, Grenoble, Rhone
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Priest-en-Jarez, Rhone
  - Hôpital Arnaud De Villeneuve - Service des Maladies Respiratoires, Montpellier
  - CHU de Nice Hôpital Pasteur - Pavillon H - Service Pneumologie, Nice
- Germany (10):
  - "Universitätsklinikum Freiburg - Medizinische Universitätsklinik, Freiburg im Breisgau, Baden-Wurttemberg
  - Thoraxklinik am Universitätsklinikum Heidelberg-Zentrum für Pulmonale Hypertension, Heidelberg, Baden-Wurttemberg
  - Waldburg-Zeil Kliniken - Fachkliniken Wangen Klinik für Pneumologie, Wangen, Baden-Wurttemberg
  - Klinikum der Universität Regensburg - Klinik und Poliklinik für Innere Medizin II, Regensburg, Bavaria
  - Medizinische Hochschule Hannover-Abteilung für Pneumologie, Hanover, Lower Saxony
  - Universitätsmedizin Greifswald Zentrum für innere Medizin Klinik und Poliklinik für Innere Medizin B, Greifswald, Mecklenburg-Vorpommern
  - Technische Universitaet Dresden - Universitaetsklinikum Carl Gustav Carus - Medizinische Klinik und Poliklinik I, Dresden, Saxony
  - Universitätsklinikum Leipzig-Dept. für Innere MedizinAbteilung für Pneumologie, Leipzig, Saxony
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - Unfallkrankenhaus Berlin-Klinik für Innere Medizin/Kardiologie, Berlin
- Israel (8):
  - Barzilai University Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Hadassah University Medical Center, Jerusalem
  - Meir Medical Center - Pulmonology Dept., Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (4):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, BG
  - Azienda Ospedaliera San Gerardo - Monza, Monza, MI
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo, PA
  - A.O.U. Policlinico Umberto I- Università La Sapienza, Roma, RM
- Vrije Universiteit Medisch Centrum (VUMC), Amsterdam, Netherlands
- Portugal (3):
  - Hospital Garcia de Orta, Almada, Lisbon District
  - Universidade de Coimbra - Hospitais da Universidade de Coimbra (H.U.C), Coimbra, Mondego
  - Centro Hospitalar de Lisboa Norte - Hospital de Santa Maria, Lisbon
- Serbia (5):
  - Clinical Center of Serbia Department of Cardiology and Polyclinic, Belgrade
  - Clinical Center of Serbia, Polyclinic, Pulomology Department, Belgrade
  - Clinical-Hospital Center Zemun, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Center of Nis, Clinic for Cardiovascular Diseases, Niš
- Spain (9):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Marques de Valdecilla (HUMV), Santander, Cantabria
  - Hospital Virgen de la Salud (HVS), Toledo, Castille-La Mancha
  - Hospital Universitario Puerta de Hierro - Madrid, Majadahonda, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Vall d'hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Valladolid, Valladolid
- Ukraine (6):
  - Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiac Surgery of Dnipropetrovsk Regional Council, Department of Cardiology, Dnipro
  - Municipal Institution of health care "Kharkiv City Clinical Hospital №13", Pulmonology Department №1, Kharkiv
  - Government Institution "L.T.Malaya Therapy National Institute of the National Academy of Medical Sciences of Ukraine", Cardiopulmonology Department, Kharkiv
  - National institute of phthisiology and pulmonology, Kyiv
  - National Scientific Centre "M.D. STRAZHESKO INSTITUTE OF CARDIOLOGY, MAS OF UKRAINE", Kyiv
  - Lviv Regional Clinical Hospital, Department of Intesive Care #2, Lviv
- United Kingdom (4):
  - Freeman Hospital, Newcastle upon Tyne, Newcastle
  - Golden Jubilee National Hospital, Clydebank, West Dunbartonshire
  - Royal Free Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants did not meet the inclusion and/or exclusion criteria and were not randomized
Groups:
- Inhaled Nitric Oxide: Randomized to Inhaled Nitric Oxide at dose of 15mcg/Kg IBW/hr for Run In Period of first 2 weeks (Week 0 and 1). Followed by Inhaled Nitric Oxide at dose of 75 mcg/kg IBW/hr for 16 weeks (Week 2 to Week 18)
- Placebo: Randomized to Placebo at dose of 15mcg/Kg IBW/hr for Run In Period of first 2 weeks (Week 0 and 1). Followed by Placebo at dose of 75 mcg/kg IBW/hr for additional 16 weeks (Week 2 to Week 16)
Period: Part 1: Blinded Tx (2 Week Run In)
Arm/Group | Inhaled Nitric Oxide | Placebo
Started | 78 | 79
Participants That Actually Received Treatment (Following randomization, there were some participants that did not start treatment during this 2 week run in period that is used to determine ability to comply with using the drug/device combination treatment therapy before they are moved to the treatment dose (75 mcg/kg IBW/hr) at Week 2.) | 74 | 78
Completed | 52 | 59
Not Completed | 26 | 20
Period: Part 1: Blinded Tx (16 Weeks)
Arm/Group | Inhaled Nitric Oxide | Placebo
Started | 52 | 58 (59 placebo subjects completed the 2 week run in period. 1 subject opted NOT to continue to the 16 week treatment period that followed and therefore, in the Blinded Tx phase there were only 58 that started.)
Completed | 40 | 42
Not Completed | 12 | 16
Period: Part 2: Open Label Extension Period
Arm/Group | Inhaled Nitric Oxide | Placebo
Started | 40 | 42
Completed ("Completed" indicates the subjects that were in Part 2 (Open Label Extension) at the time of the Interim Analysis when the study was early terminated for futility.) | 40 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis set includes all randomized subjects who remained eligible after 2 week run in period (dose 15 mcg/kg IBW/hr) that wanted to continue into treatment period of 16 weeks at study dose (75 mcg/kg IBW/hr)
Groups:
- Inhaled Nitric Oxide: Includes all randomized subjects that completed 2 week run in period and opted to continue with 16 week treatment period. Treated with Inhaled Nitric Oxide at dose of 75 mcg/Kg IBW/hr
- Placebo: Includes all randomized subjects that completed 2 week run in period and opted to continue with 16 week treatment period. Treated with Placebo at dose of 75 mcg/Kg IBW/hr
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Placebo | Total
Number analyzed (Participants) | 52 | 58 | 110
Age, Continuous [Median (Full Range); unit: Years] | 65 [22 to 81] | 63 [26 to 80] | 64 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 12 | 22 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 51 | 56 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 52 | 55 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
6 Minute Walk Distance (6MWD) [Median (Full Range); unit: meters] | 286 [80 to 476] | 323 [117 to 555] | 312 [80 to 555]
Oxygen Use (Hours/Day) at Baseline [Count of Participants; unit: Participants]
  <8 hours per day | 46 | 49 | 95
  >8 hours per day | 6 | 9 | 15
Cardiac Index [Median (Full Range); unit: L/minute/m^2] — Baseline considered Day of Randomization (Day 0).
  Reported as Derived Cardiac Index (CI) where Derived CI = Cardiac Output (CO) / BSA. Where Patient's BSA (Body Surface Area) = 0.007184*(weight^0.425)*(Height^0.725).
  All pulmonary hemodynamic measurements including CO used in the derived CI measured from Right Heart Catheterization (RHC) collected at Baseline (Day of Randomization).
  L/minute/m^2 | 2.05 [1.6 to 3.5] | 2.30 [1.9 to 2.7] | 2.18 [1.6 to 3.5]
Pulmonary Vascular Resistance (PVR) via RHC [Median (Full Range); unit: dynes.second/cm^5] — Baseline considered Day of Randomization (Day 0).
  Pulmonary Vascular Resistance (PVR) measured from Right Heart Catheterization (RHC) collected at Baseline (Day of Randomization).
  dynes.second/cm^5 | 726 [276 to 2080] | 940 [413 to 1147] | 839 [276 to 2080]

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Distance (6MWD) From Baseline (Randomization) to End of Treatment Period (Week 18)
Description: The 6-minute walk distance test (6MWD) is a non-encouraged test performed in a 30 m long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. All patients were required to complete two walks while on chronic oxygen therapy given at a standard rate during the test and throughout the study while using the investigational product (INOpulse device with nitric oxide or matching placebo). The average of two walks at Week 2 visit (2 weeks after Run-In) was used as the Baseline 6MWD.
Time Frame: Change in 6MWD from Week 2 (2 weeks after randomization and run-in period) to Week 18 (end of blinded treatment period)
Population: 6MWD Change from Week 2 (2 weeks after randomization and run-in period) to Week 18 (end of blinded treatment period) (Week 18). MMRM model includes Baseline 6MWD as covariate, Treatment Group, Visit, Prostanoids usage status and Treatment by Visit Interaction as fixed effects. No imputation performed for primary analysis. ITT analysis set only includes study participants that completed 16 weeks of Part 1 blinded treatment.
Measure: Least Squares Mean (Standard Error); unit: meters
Groups:
- Inhaled Nitric Oxide 75mcg/KgIBW/Hr: Part 1: Blinded Treatment - 75 mcg/Kg IBW/hr for 16 weeks (included only participants who were compliant in the first 2 weeks)
- Placebo: Part 1 Blinded Treatment - Placebo dose setting 75 mcg/kg IBW/hr for 16 weeks (included only participants who were compliant in the first 2 weeks)
Arm/Group | Inhaled Nitric Oxide 75mcg/KgIBW/Hr | Placebo
Number analyzed (Participants) | 52 | 58
meters | 4.88 (6.90) | 2.89 (10.13)
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide 75mcg/KgIBW/Hr vs Placebo; Test type: Superiority; p = 0.87, Mixed Models Analysis; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [-22.47 to 26.45]

2. Secondary Outcome: Time (in Days) to First Clinical Worsening Event (TTCW)
Description: Clinical worsening was assessed continuously from Randomization to Week 18 (End of blinded treatment period). Clinical worsening events were defined as death (all causes), atrial septostomy, hospitalization due to worsening of pulmonary arterial hypertension (PAH), initiation of new pulmonary arterial hypertension treatment including endothelin receptor antagonists [ERAs], phosphodiesterase type-5 [PDE-5] inhibitors or prostanoids, an increase in existing treatment of ERA or PDE-5, increase in the dose or frequency of an inhaled prostanoids, or an increase in the dose of an intravenous or subcutaneous prostanoids by >10%, a decrease of >15% from baseline or >30% compared with the last study related measurement in 6MWD or worsening of WHO Functional Class (e.g., from Class II to Class III or IV, OR Class III to Class IV). All worsening events were entered by the study sites into the eCRF.
Time Frame: From Randomization to Week 18 (End of blinded treatment period)
Population: ITT analysis population
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Inhaled Nitric Oxide 75mcg/KgIBW/Hr: Part 1:
  Blinded Treatment - 15 mcg/kg IBW/hr for first 2 weeks Blinded Treatment - 75 mcg/Kg IBW/hr for 16 weeks (included only participants who were compliant in the first 2 weeks)
- Placebo: Part 1:
  Blinded Treatment - Placebo dose setting 15mcg/kg IBW/hr for first 2 weeks Blinded Treatment - Placebo dose setting 75 mcg/kg IBW/hr for 16 weeks (included only participants who were compliant in the first 2 weeks)
Arm/Group | Inhaled Nitric Oxide 75mcg/KgIBW/Hr | Placebo
Number analyzed (Participants) | 52 | 58
Days | 22 (42.3) | 19 (32.8)
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide 75mcg/KgIBW/Hr vs Placebo; Test type: Superiority; p = 0.55, Log Rank

3. Secondary Outcome: Number of Participants With an Improvement in World Health Organization Functional Class (WHO FC) Baseline (Randomization) to End of Treatment Period (Week 18)
Description: WHO FC (where Class I is defined as "No limitations in daily physical activities. No symptoms of dyspnea and with routine exertion" and Class IV is defined as "Inability to perform even minimal activities. Signs and symptoms of right heart failure may be present. Dyspnea present at rest") for PAH was taken at randomization (Week 0) for all participants and was assessed after blinded treatment (Week 18). The number of participants that had an improvement (lower functional class) as compared to baseline were measured.
Time Frame: From Randomization to Week 18 (End of blinded treatment period)
Population: ITT analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide 75mcg/KgIBW/Hr | Placebo
Number analyzed (Participants) | 52 | 58
Participants | 2 | 1

4. Other Pre Specified Outcome: Change in Plasma N-Terminal Pro-brain Natriuretic Peptide (NT-proBNP) From Screening to End of Treatment Period (Week 18)
Description: Plasma NT-proBNP concentration is a useful biomarker for the severity of PAH as it is associated with changes in right heart morphology and function. NT-proBNP sample collection occurred at Screening visit (prior to starting study drug at Randomization) and after 16 weeks of blinded treatment therapy (Week 18). The change in NT-proBNP between Screening (28 days prior to baseline/randomization) and the end of blinded treatment period (Week 18) is reported.
Time Frame: From Screening (28 days prior to baseline/randomization) to end of Blinded Treatment Period (Week 18)
Population: ITT analysis population who had NT Pro BNP levels at Screening and at the end of blinded treatment period (Week 18)
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Inhaled Nitric Oxide 75mcg/KgIBW/Hr | Placebo
Number analyzed (Participants) | 34 | 30
pg/mL | 117.8 (22.8) | 207.9 (24.8)
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide 75mcg/KgIBW/Hr vs Placebo; Test type: Superiority; p = 0.01, ANCOVA; Mean Difference (Final Values) = -89.1, 95% CI 2-sided [-156.0 to -22.1]

5. Other Pre Specified Outcome: Change in Borg Dyspnea Scale Immediately Following 6-minute Walk Test (6MWT) From Baseline (Randomization) to End of Treatment Period (Week 18)
Description: The Borg dyspneas score is a self-rating scale to evaluate the severity of dyspnea (from 0 "no shortness of breath at all" to 10 "very, very severe / maximal") shortness of breath, where high score on the scale signifies a worse score. The self assessment was collected from each participant immediately after each 6-minute walk test throughout the blinded treatment period. The change in Borg dyspnea Score at the end of the blinded treatment period (Week 18) compared to baseline (randomization) (Week 0) is reported.
Time Frame: From Randomization to Week 18 (End of blinded treatment period)
Population: ITT analysis population
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Inhaled Nitric Oxide 75mcg/KgIBW/Hr | Placebo
Number analyzed (Participants) | 52 | 58
Scores on a Scale | -0.47 (0.23) | -0.23 (0.23)
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide 75mcg/KgIBW/Hr vs Placebo; Test type: Superiority; p = 0.47, ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.89 to 0.41]

6. Other Pre Specified Outcome: Number of Participants With an Unsatisfactory Clinical Response From Baseline (Randomization) to End of Treatment Period (Week 18)
Description: Unsatisfactory Clinical Response was defined as the number of participants with WHO Functional Class III (defined as moderate dyspnea with routine activities and activities of daily living. No symptoms at rest.) or Class IV (defined as inability to perform even minimal activities. Signs and symptoms of right heart failure may be present. Dyspnea present at rest) with no improvement in 6-minute walk distance (6MWD) from baseline to end of blinded treatment period (Week 18).
Time Frame: From Randomization to Week 18 (End of blinded treatment period)
Population: ITT analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide 75mcg/KgIBW/Hr | Placebo
Number analyzed (Participants) | 52 | 58
Participants | 32 | 35
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide 75mcg/KgIBW/Hr vs Placebo; Test type: Superiority; p = 0.26, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.48 to 2.29]

ADVERSE EVENTS:
Time Frame: Adverse events data collected from all participants that were enrolled in the study and who actually received study treatment in Part 1 (up to 18 weeks) and in Part 2 (up to 30 weeks).
Description: Note that adverse events are presented together for Parts 1 (Run-in, Treatment) and 2 (Open label). Adverse events were not monitored/assessed separately for the Run-in (2 week), Blinded Treatment (16 week) period (Part 1) and Open Label (Part 2) periods. The Number of Participants At-Risk includes participants from both Parts 1 and 2.
Groups:
- Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Inhaled Nitric Oxide and Part 2 - Inhaled Nitric Oxide: Part 1 Randomized to Inhaled Nitric Oxide that was actually treated at dose of 15mcg/Kg IBW/hr for Run In Period of first 2 weeks (Week 0 and 1).
  Followed by Inhaled Nitric Oxide at dose of 75 mcg/kg IBW/hr for 16 weeks (Week 2 to Week 18)
  Part 2 Following by open label treatment with Inhaled Nitric Oxide
- Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Placebo and Part 2 - Placebo: Randomized to Placebo that was actually treated at at dose of 15mcg/Kg IBW/hr for Run In Period of first 2 weeks (Week 0 and 1).
  Followed by placebo at dose of 75 mcg/kg IBW/hr for 16 weeks (Week 2 to Week 18)
  Part 2 Following by open label treatment with Inhaled Nitric Oxide
Arm/Group | Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Inhaled Nitric Oxide and Part 2 - Inhaled Nitric Oxide | Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Placebo and Part 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 2/74 | 3/78
Serious Adverse Events (participants affected / at risk) | 13/74 | 10/78
Other Adverse Events (participants affected / at risk) | 22/74 | 25/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Inhaled Nitric Oxide and Part 2 - Inhaled Nitric Oxide (N=74) | Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Placebo and Part 2 - Placebo (N=78)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Presyncope (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung transplant (Surgical and medical procedures) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Inhaled Nitric Oxide and Part 2 - Inhaled Nitric Oxide (N=74) | Part 1:Blinded Tx (2 Week Run In & 16 Weeks) Placebo and Part 2 - Placebo (N=78)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 3 | 4
Cardiac failure (Cardiac disorders) | 0 | 2
Oedema peripheral (Cardiac disorders) | 2 | 1
Presyncope (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute right ventricular failure (Cardiac disorders) | 1 | 0
Acute right ventricular failure (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Chest pain (Cardiac disorders) | 1 | 0
Fluid overload (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eye infection (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Asthenia (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Secretion discharge (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Drug ineffective (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Influenza (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 0 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 1
Right ventricular ejection fraction decreased (Investigations) | 1 | 0
Serum ferritin decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Device failure (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 3 | 1
Ecchymosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Planned Interim Analysis resulted in early termination due to futility, leading to small numbers of study participants analyzed. Analysis is based on Part 1 Blinded Treatment Period (up to 18 Weeks) only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02725372/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT02725372/SAP_001.pdf